CLINICAL TRIAL: NCT07400224
Title: Clinical Application of Al18F-NOTA-FAPI-04 PET/CT or PET/MRI Imaging in Malignant Tumor,Cardiovascular or Immune Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JS-3423
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Hyperthyroidism, Autoimmune; Cardiovascular Abnormalities; Malignant Tumor
MeSH Terms: conditions — Graves Disease; Cardiovascular Abnormalities; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-NOTA-FAPI PET/CT(PET/MRI) (Experimental): Evaluation of dosimetry, safety, diagnostic accuracy, and clinical treatment strategy guidance ability of Al18F-NOTA-FAPI PET/CT(or PET/MRI) in patients with malignant tumor,cardiovascular or immune disease.
  Interventions: Other: Al18F-NOTA-FAPI PET/CT(or PET/MRI)

INTERVENTIONS:
Other: Al18F-NOTA-FAPI PET/CT(or PET/MRI) — Participants will receive an intravenous injection of Al18F-NOTA-FAPI, prepared on-site and measured by qualified personnel using a dose calibrator, with readings and time recorded. The radiopharmaceutical will be slowly administered through a three-way stopcock, followed by a flush with 5 mL of normal saline. The recommended dose is approximately 4.81 MBq/kg (0.13 mCi/kg) body weight, with variations depending on drug yield and clinical scheduling. PET/CT(or PET/MRI) imaging are planned 45-90 minutes after administration, with adjustments based on drug yield and equipment availability.

SUMMARY:
This prospective, single-center study investigates the biodistribution, dosimetry, safety, diagnostic performance of Al18F-NOTA-FAPI PET imaging in patients with malignant tumor,cardiovascular or immune disease. And evaluates the potential of Al18F-NOTA-FAPI PET imaging in Clinical treatment strategy guidance.

DETAILED DESCRIPTION:
FAP is expected to become an important indicator for predicting tumor prognosis, and also a new target for individualized treatment of various diseases such as tumors, rheumatoid arthritis, myocardial infarction, and thyroid-associated ophthalmopathy. The biological distribution of FAP in healthy adults is not yet clear. It is planned to obtain the normal PET/CT (or PET/MRI) images of healthy subjects after they use this tracer, in order to establish a benchmark for future application in patients.

ELIGIBILITY:
Inclusion Criteria:

* a. Age 18 years old or above, gender not restricted. b. Have undergone a health check-up within the last 3 months (at least completed chest X-ray / chest CT and abdominal B-ultrasound and other examinations), and no major diseases were found.

Exclusion Criteria:

* As this study involves certain radiation exposure, patients who have had frequent radiation exposure due to clinical needs (those who have undergone a CT or PET/CT examination once within 3 months or 1 month respectively) are not included in the study.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Al18F-NOTA-FAPI | From radiotracer injection to 24 hours post-injection.
  Adverse effects were recorded according to CTCAE (version 5.0) after radiotracer injection and PET scan.
Diagnostic accuracy of Al18F-NOTA-FAPI PET/CT(PET/MRI) for cardiovascular or immune disease. | Through study completion, 1-1.5 years .
  SUVmax 、SUVmean and T2 value（MRI）of the heart and the eye muscles will be measured. Two nuclear medicine physicians will independently review the images, and a third physician will adjudicate in case of disagreement to reach a final diagnosis. Surgical pathology results or Long term follow up findings will serve as the reference standard to determine the sensitivity and specificity .

SECONDARY OUTCOMES:
SUVmax of normal organs | From study completion to 6 months after completion.
  The biodistribution of Al18F-NOTA-FAPI will be assessed in the following organs: pituitary gland, parotid glands, thyroid glands, lungs, blood pool, liver, spleen, pancreas (including the head and uncinate process), gallbladder, stomach, small intestine, kidneys, and adrenal glands. The SUVmax values for these organs will be measured and documented.
Absorbed dose of target organs | From study completion to 6 months after completion
  Absorbed dose of target organs were calculated using HERMES software.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided